CLINICAL TRIAL: NCT02460172
Title: A Prospective, Randomized Controlled Post-market Study to Compare the Use of the Zip® Surgical Skin Closure Device Versus Conventional Staples for Skin Closure in Subjects Having Undergone Bilateral Knee Arthroplasty
Brief Title: Zip® Surgical Skin Closure Device vs. Staples for Skin Closure in Subjects Having Undergone Bilateral Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ZipLine Medical Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 006
Record Dates: First submitted 2015-05-28; First posted 2015-06-02 (Estimated); Results first posted 2019-03-05 (Actual); Last update posted 2019-03-05 (Actual); Status verified 2019-02

CONDITIONS: Arthroplasty, Knee Replacement; Wound Healing
Keywords: bi lateral; knee surgery; arthroplasty; orthopedics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Zip Surgical Skin Closure (Active Comparator): Subject will be randomized to receive one knee (right or left) closed with Zip Surgical Skin Closure and the other knee closed with steel staples.
  Interventions: Device: Zip Surgical Skin Closure
- Steel Staples (Active Comparator): Subject will be randomized to receive one knee (right or left) closed with steel staples and the other knee closed with Zip Surgical Skin Closure.
  Interventions: Device: Steel Staples

INTERVENTIONS:
Device: Zip Surgical Skin Closure — Non invasive, reversible, skin closure device for closure of the skin layer following surgical incisions or laceration repair.
  Other Names: Zip16; Zip 8i
  Arms: Zip Surgical Skin Closure
Device: Steel Staples — Skin closure device for the closure of the skin layer following surgical incision
  Other Names: Conventional staples
  Arms: Steel Staples

SUMMARY:
Study designed to compare the Zip Surgical Skin Closure device vs. conventional staples for wound closure following bi lateral knee replacement surgery.

DETAILED DESCRIPTION:
Prospective, randomized, within patient control study comparing the use of Zip Surgical Skin Closure device versus conventional staple placement when utilized for surgical wound closure after bi lateral unicompartmental or bi lateral total knee replacement. A total of up to 25 patients will be enrolled and followed for up to 8 weeks post surgery to evaluate wound healing and overall satisfaction of closure method.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 18 years of age and older
2. Patients requiring epidermal closure after bi lateral total or partial (unicompartmental) knee arthroplasty
3. Patients willing to be evaluated at discharge, 2 weeks, and at the 6 to 8 week post op

Exclusion Criteria:

1. Known bleeding disorder not caused by medication
2. Known personal or family history of keloid formation or scar hypertrophy
3. Known allergy or hypersensitivity to non-latex skin adhesives
4. Atrophic skin deemed clinically prone to blistering
5. Any skin disorder affecting wound healing
6. Any other condition that in the opinion of the investigator would make a particular patient unsuitable for this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2017-02-15 (Actual); Study Completion 2017-02-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rodney Benner, MD, Principal Investigator — Study Center
Locations (1):
- Shelbourne Knee Center, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is a split person study where one knee is assigned Zip, the other knee is assigned Staples. 50 knees were closed on 25 participants.
Units Other Than Participants: knees
Groups:
- All Participants: Subject will be randomized to receive one knee (right or left) closed with steel staples and the other knee closed with Zip Surgical Skin Closure.
  Zip Surgical Skin Closure: Non invasive, reversible, skin closure device for closure of the skin layer following surgical incisions or laceration repair.
  Steel Staples: Skin closure device for the closure of the skin layer following surgical incision.
Period: Overall Study
Arm/Group | All Participants
Started (This is a split-person study) | 25; 50 knees
Completed | 25; 50 knees
Not Completed | 0; 0 knees

BASELINE CHARACTERISTICS:
Population: Patients requiring epidermal closure after bi lateral total or partial (unicompartmental) knee arthroplasty
Groups:
- All Participants: Subject will be randomized to receive one knee (right or left) closed with Zip Surgical Skin Closure and the other knee closed with steel staples.
  Zip Surgical Skin Closure: Non invasive, reversible, skin closure device for closure of the skin layer following surgical incisions or laceration repair.
  Steel Staples: Skin closure device for the closure of the skin layer following surgical incision.
Arm/Group | All Participants
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.7 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 13
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 23
  Black/African Amer. | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 25
Range of Motion [Mean (Standard Deviation); unit: degrees] — Range of Motion for each knee will be measured (Left and Right)
  degrees
    Knees assigned Zip closure | 121 (13.66)
    Knees assigned Staple closure | 118 (25.99)

OUTCOME MEASURES:

1. Primary Outcome: Incision Appearance / Scar Cosmesis
Description: Patient Scar Rating (0=Best to 10=Worst). A lower score means better scar rating.
  Surgeon Scar Rating (0=Best to 10=Worst). A lower score means better scar rating.
  Independent Plastic Surgeon Scar Rating by 8 week post op photos. (0=Best to 10=Worst). A lower score means better scar rating.
Time Frame: 6-8 weeks post surgery
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Zip Surgical Skin Closure: Subject will be randomized to receive one knee (right or left) closed with Zip Surgical Skin Closure and the other knee closed with steel staples.
  Zip Surgical Skin Closure: Non invasive, reversible, skin closure device for closure of the skin layer following surgical incisions or laceration repair.
  Steel Staples: Skin closure device for the closure of the skin layer following surgical incision.
- Steel Staples: Subject will be randomized to receive one knee (right or left) closed with steel staples and the other knee closed with Zip Surgical Skin Closure.
  Zip Surgical Skin Closure: Non invasive, reversible, skin closure device for closure of the skin layer following surgical incisions or laceration repair.
  Steel Staples: Skin closure device for the closure of the skin layer following surgical incision.
Arm/Group | Zip Surgical Skin Closure | Steel Staples
Number analyzed (Participants) | 25 | 25
units on a scale
  Patient Rating | 1.3 (0.5) | 2.6 (2.4)
  Surgeon Rating | 1.9 (1.2) | 3.3 (1.0)
  Plastic Surgeon Rating | 3.7 (2.0) | 4.8 (1.8)

2. Secondary Outcome: Surgeon Closure Method Satisfaction
Description: Closure method satisfaction will be collected by a 5 point satisfaction scale:
  1. Very Satisfied
  2. Satisfied
  3. Neither
  4. Dissatisfied
  5. Very Dissatisfied A lower score means more satisfaction with the closure method.
Time Frame: 6-8 weeks post op
Measure: Count of Participants; unit: Participants
Arm/Group | Zip Surgical Skin Closure | Steel Staples
Number analyzed (Participants) | 25 | 25
Participants
  Surgeon Very Satisfied | 17 | 5
  Surgeon Satisfied | 7 | 17
  Surgeon Neither Satisfied or Dissatisfied | 1 | 3

3. Secondary Outcome: Patient Pain - Incisional and General
Description: Pain levels will be collected using a 10 point VAS scale.
Time Frame: Throughout 8 week study period (Discharge, 2 wk follow up and 8 wk exit visit)
Population: Patient incisional pain scores for Zip side and incisional pain scores for Staples side were collected (0=no pain, 10=worst pain imaginable)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Zip Surgical Skin Closure | Steel Staples
Number analyzed (Participants) | 25 | 25
units on a scale
  Discharge Pain | 1.8 (2.0) | 2.4 (2.6)
  2 Week Pain pre removal | 1.4 (1.7) | 2.0 (1.8)
  2 Week Pain post removal | 0.7 (1.1) | 1.6 (1.2)
  6 to 8 Week Pain | 0.5 (0.1) | 0.9 (1.4)

4. Secondary Outcome: Surgeon and Patient Scar Satisfaction
Description: Scar Satisfaction (both Zip and Staple sides) will be collected using a 5 point scale:
  Very Satisfied Satisfied Neither Dissatisfied Very Dissatisfied
Time Frame: 6 to 8 wk follow up visit
Measure: Count of Participants; unit: Participants
Arm/Group | Zip Surgical Skin Closure | Steel Staples
Number analyzed (Participants) | 25 | 25
Participants
  Surgeon Scar Satisfaction: Very Satisfied | 17 | 5
  Surgeon Scar Satisfaction: Satisfied | 7 | 17
  Surgeon Scar Satisfaction: Neither | 1 | 3
  Surgeon Scar Satisfaction: Dissatisfied | 0 | 0
  Surgeon Scar Satisfaction: Very Dissatisfied | 0 | 0
  Patient Scar Satisfaction: Very Satisfied | 18 | 8
  Patient Scar Satisfaction: Satisfied | 4 | 7
  Patient Scar Satisfaction: Neither | 3 | 7
  Patient Scar Satisfaction: Dissatisfied | 0 | 3
  Patient Scar Satisfaction: Very Dissatisfied | 0 | 0

5. Secondary Outcome: Range of Motion
Description: Knee Range of Motion for each knee will be measured in degrees
Time Frame: 2 weeks and 6-8 weeks
Measure: Mean (Standard Deviation); unit: degrees
Units Other Than Participants: knees
Arm/Group | Zip Surgical Skin Closure | Steel Staples
Number analyzed (Participants) | 25 | 25
Number analyzed (knees) | 25 | 25
degrees
  2 week Range of Motion | 109 (11.79) | 105 (13.64)
  6-8 Week Range of Motion | 122 (10.78) | 122 (10.82)

ADVERSE EVENTS:
Time Frame: Up to Study Exit at 6 to 8 Week Follow Up
Description: No Serious Adverse Events No All Cause Mortality
Arm/Group | Zip Surgical Skin Closure | Steel Staples
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 1/25 | 0/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zip Surgical Skin Closure (N=25) | Steel Staples (N=25)
Superficial Skin Peeling (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Superficial skin peeling upon device removal

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-04-21): https://cdn.clinicaltrials.gov/large-docs/72/NCT02460172/Prot_SAP_000.pdf